CLINICAL TRIAL: NCT06235177
Title: Psychoneuromentalism Disorder: A Condition Resulting From Behavioral Impairments, Neurodiversity, and Neurobehavioral Dysfunctions Related to the Mental and Emotional State of a Person
Brief Title: Psychoneuromentalism Disorder: A Medical Condition That Affects People With Psychological Impairments From Health Issues
Acronym: PNMD
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Essence of Integrative Health and Medicine Practice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EssenceIntegrativeHlth
Record Dates: First submitted 2021-12-13; First posted 2024-01-31 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Schizoaffective Disorder, Bipolar Type; Bipolar Disorder; ADHD - Combined Type; Dissociative Disorder; Stress Disorder; Dementia; Anxiety; Chronic Fatigue Syndrome
Keywords: Psychology; Neuroscience; Mental Health; Disorder; Stress; Anxiety; Psychoneuromentalism Disorder; ADHD; Fatigue
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Dissociative Disorders; Stress Disorders, Traumatic; Dementia; Anxiety Disorders; Fatigue Syndrome, Chronic; Psychological Well-Being; Disease; Attention Deficit Disorder with Hyperactivity; Fatigue | interventions — Mindfulness; Dietary Supplements; Vitamins; Meditation; Breathing Exercises; Music Therapy

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to find individuals who do not have a primary psychological disorder prior to a medical condition, behavior change, or a shift in the mind and body from a traumatic experience, PTSD, Dementia, Stress, and physical limitations that has caused a psychological issue.The other purpose is to assist the participants in naturopathy/holistic medicine treatments, which will allow them to not only recover from their current condition, but to also have an overall well-being, become more sustainable in their daily lives, and have an overall sense of health.
Masking Description: Recent studies suggest that neurotrophic factors play an important role in the pathogenesis of depression as well as the therapies for depression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Techniques for Psychoneuromentalism Disorder (Experimental): The Interventions to be administered will be as follows:
  1. Ashwagandha Herb Tincture and Supplement
  2. Damiana Herb Tincture
  3. Passion Flower Herb Tincture
  4. Grapeseed Extract- Capsule
  5. Rhodiola- Herb Tincture
  6. Sea Moss Supplement Capsule
  7. Theocentric Psychological Counseling
  8. Clinical Yoga
  9. Meditation
  10. Mental Imagery
  11. Decompartmentalization Framework
  12. Dietary Supplements
  13. Applied Relaxation (Music Meditation, Breathing Techniques)
  14. Pain Relaxation Techniques
  15. Meridian Acupuncture
  Interventions: Combination Product: Decompartmentalization Framework; Dietary Supplement: Liquid Herbal TInctures; Other: Mental Imagery; Diagnostic Test: Clinical Yoga; Dietary Supplement: Dietary Supplements; Behavioral: Applied Relaxation; Behavioral: Pain Relaxation Techniques; Behavioral: Comprehensive Theocentric Psychological Assessment

INTERVENTIONS:
Combination Product: Decompartmentalization Framework — I will also be using mental imagery, consciousness, cognition, and cognitive psychology during this study to show the effectiveness of the conscious mind, and how the mind can influence behavior.
  Decompartmentalize means to remove excessive compartmentalization; to restore from a compartmentalized state; to merge back together.
Dietary Supplement: Liquid Herbal TInctures — I will make and administer liquid herbal tinctures that will be made from all natural leafs, roots and flowers. I will focus on and track the participants' diagnosis, side effects, and how they feel before, during and after taking the liquid tincture.
  Other Names: Herbal Tincture
Other: Mental Imagery — I will have the participants focus on a particular shape, sound or image that they can see, think, or hear. This will allow the participant to have a clear mind, and release any negative thoughts, negative energy and boost their moods and their 5 senses.
  Other Names: Mindfulness
Diagnostic Test: Clinical Yoga — I will show the participants many different yoga positions that will give them a peace of mind, stretch their muscles and release any tension throughout their body, and have an overall well-being, as well as promoting mindfulness.
  Other Names: Yoga, Mediation
Dietary Supplement: Dietary Supplements — I will have the participants take an herbal supplement and/or vitamin that relates to the symptoms and current issues/diagnosis they have. The Dietary Supplements/Vitamins will enhance their capacity to overcome their health conditions, protect their body from unwanted germs and bacteria, and relieve the participants' mind and body from the symptoms they are experiencing based on their current condition.
  Other Names: Vitamins
Behavioral: Applied Relaxation — Applied Relaxation is a specialized form of relaxation training that aims to teach the participant how to relax in common social situations.
  Mindfulness training encourages participants to gain psychological distance from their worries and negative emotions, seeing them as an observer would see them. 2 types of mindfulness will be used, which is mindfulness-based stress reduction and mindfulness-based cognitive therapy. Treatment starts with general education about stress and social anxiety.
  Other Names: Meditation, Breathing Exercises, Music Therapy
Behavioral: Pain Relaxation Techniques — Relaxation can reduce the feelings of stress, helping them to gain more control. Reduce pain by decreasing muscle tension, aches and pains. The body releases endorphins (the body's natural pain-killers) to relieve pain.
  Yoga incorporates breath control, meditation, and gentle movements to stretch and strengthen muscles.
  Mind-body techniques, which includes meditation, mindfulness, and breathing exercises help you restore a sense of control over your body and turn down the "fight or flight" response, which can worsen chronic muscle tension and pain.
Behavioral: Comprehensive Theocentric Psychological Assessment — To enhance the lives of add to the lives of those who are well adjusted but know they have a greater potential within themselves to ring forth and live more fulfilling lives,

SUMMARY:
Psychoneuromentalism Disorder is a disorder arising in the mind; that is related to the mental and emotional state of a person. It is the science of mental life. The body has a natural design to heal itself. This is a mental phenomena that cannot be explained, until now.

Psychoneuromentalism Disorder is a new condition resulting from behavioral impairments, neurodiversity, and neurobehavioral dysfunctions that are related to the mental and emotional state of a participant.

DETAILED DESCRIPTION:
To further explain this new medical condition that I created, I'd like to break down the components of Psychoneuromentalism Disorder.

Mentalism is the theory that physical and psychological phenomena are explicable only in terms of a creative and interpretative mind; which means it relies on pure belief. These are the branches of study that concentrate on perception and thought processes. There is a psychological theory that states that humans possess a conscious mind, and that the mind can influence behavior.

Conscious means that a person is aware of their surroundings, having knowledge of something, sensitive to their inner realization of a fact, truth, or condition. A behavioral approach suggests that the keys to understanding development are observable behavior and external stimuli in the environment--- it is a theory of learning, and learning theories that focus on how we are conditioned to respond to events or stimuli. Mentalism is also the doctrine that the mind is the fundamental reality and that objects of knowledge exist only as aspects of the participants consciousness.

Disorder is a functional abnormality or disturbance. It is an illness that disrupts the normal physical or mental functions. It is a set of problems, which result in causing significant difficulty, distress, impairment, and/or suffering in a participants daily life.

Neuroscience focuses on the brain and its impact on the behavior and cognitive functions. It is concerned with the normal functioning of the nervous system, and what also happens to the nervous system when people have neurological, psychiatric, and neurodevelopmental disorders.

Neurobehavioral difficulties include 2 primary categories:

1. Cognitive decline, including memory problems, and dementia, and
2. neuropsychiatric disorders, including neurasthenia (difficulty concentrating, headache, insomnia, and fatigue), depression, post-traumatic stress disorder and suicide.

There have always been neurodevelopmental disturbances that refers to variations in the brain regarding sociability, learning, attention, mood, and other mental functions. ADHD, developmental speech disorders, dyslexia, dyspraxia, dyscalculia, dyssomnia, intellectual disability, and Mental health conditions such as bipolar disorder, schizophrenia, schizoaffective disorder, antisocial personality disorder, disassociated disorders, OCD, Stress, and localized anxiety disorders. Neurodiversity advocates point out that neuro-diverse people often have exceptional abilities such as hyper-focus alongside their deficits.

Hyper-focus is an intense fixation on an interest or activity for an extended period of time, and most participants block out the world around them. Therefore, the brain is less sensitive to the chemical; dopamine, which is linked to reward and attention, which is what most participants are looking for.

The body has a natural design to heal itself. It is deep and intense concentration. Psychoneuromentalism Disorder is a disorder arising in the mind; that is related to the mental and emotional state of a person. It is the science of mental life. The body has a natural design to heal itself. This is a mental phenomena that cannot be explained, until now.

Psychoneuromentalism Disorder is a new condition resulting from behavioral impairments, neuro-diversity, and neuro-behavioral dysfunctions that are related to the mental and emotional state of a participant.

Recent studies suggest that neuro-trophic factors play an important role in the patho-genesis of depression as well as the therapies for depression. Among one of the most widely spread neuro-trophic factors in the brains of adults, is brain-derived neuro-trophic factor (BDNF), which is over-expressed in the hippocampus as well as the cerebral cortex.

Understanding Psychoneuromentalism Disorder: A Holistic Approach to Mind-Body Integration

In the realm of healthcare, the mind-body connection has long been recognized as a vital component of overall well-being. However, traditional approaches often focus solely on either mental or physical health. Enter psychoneuromentalism disorder (PNMD), a groundbreaking framework that aims to bridge this gap by considering the interconnectedness of the mind and body. Developed during my time in naturopathic medical school, PNMD seeks to address the physical ailments that can contribute to psychological distress, such as depression and stress. This article will delve into the concept of PNMD, its potential implications, and the benefits of adopting a holistic approach.

Understanding Psychoneuromentalism Disorder:

Psychoneuromentalism disorder (PNMD) is a unique medical condition that challenges the conventional view of mental illness and physical ailments as separate entities. It emphasizes the integration of the mind and body, acknowledging that psychological distress can be influenced by underlying physical imbalances and vice versa. This holistic approach recognizes that mental well-being is not solely dependent on one's thoughts and emotional state, but also on the state of one's physical health.

The Importance of Mind-Body Integration:

By considering the interplay between the mind and body, PNMD offers a more comprehensive understanding of health and illness. Stress, for instance, can manifest as physical symptoms like muscle tension, headaches, or digestive issues. Similarly, physical ailments, such as chronic pain or hormonal imbalances, can significantly impact mental well-being, leading to depression, anxiety, or other psychological disturbances. PNMD encourages healthcare professionals to explore these interconnected factors to develop more effective treatment plans.

Significance in Holistic Healthcare:

The emergence of PNMD has significant implications for the field of holistic healthcare. By adopting this framework, practitioners can provide patients with a more comprehensive and personalized approach to treatment. Rather than solely focusing on symptomatic relief or medication, PNMD encourages a multi-faceted approach that incorporates lifestyle changes, nutritional interventions, stress management techniques, and mind-body therapies. This holistic perspective empowers individuals to address the root causes of their distress and promotes overall well-being.

Benefits of PNMD:

1. Comprehensive Treatment: PNMD enables healthcare professionals to address both the physical and psychological aspects of a patient's condition, resulting in a more comprehensive and effective treatment plan.
2. Personalized Care: By recognizing the unique interplay between the mind and body, PNMD facilitates personalized care, tailoring treatment strategies to each individual's specific needs.
3. Preventive Focus: PNMD emphasizes the importance of preventive measures, encouraging individuals to proactively manage their health and well-being, thereby reducing the risk of developing chronic conditions.
4. Empowerment and Self-Care: PNMD empowers individuals to take an active role in their healthcare journey. By promoting self-care practices, patients can develop a deeper understanding of their well-being and actively participate in their own healing process.

Psychoneuromentalism disorder (PNMD) represents a paradigm shift in the way we approach mental and physical health. By acknowledging the intricate connection between the mind and body, this framework offers a more holistic understanding of health and illness. Healthcare professionals embracing PNMD can provide comprehensive, personalized care and empower individuals to achieve optimal well-being. As the field of medicine evolves, incorporating the principles of PNMD may pave the way for more effective, integrative approaches to healthcare.

Anxiety, including generalized anxiety, panic, post-traumatic stress, obsessive-compulsive, and phobic disorders is one of the principal symptoms of diverse mental disorders. The mechanism of action of anxiety disorders remain unclear.

Our mind creates our perceptions, our illusions, and our realities Our mind is reflected in our thoughts, beliefs, and attitudes. Our world is a reflection of our mind (Pert 147). It has been said that we only use one tenth of our total mental capacity. Our mind makes the landscape of our inner world. It paints scenes of thoughts, dreams, experiences, and images. The mind is responsible for feelings of joy or pain. The many aspects of our mind (attitudes, mental attributes, skills, memories, personality, and beliefs), all provide the constellation of who we are. William James stated: "Man is made or unmade by himself; in the armory of thought he forges the weapons by which he destroys himself; he also fashions the tools with which he builds for himself heavenly mansions of joy, strength, and peace" (5).

For most of us, the mind is thought to reside solely in the brain but recent research is changing our understanding. It has been found that mind is not found at any single point in our body; mind activity is now seen as much a function of body as a function of the brain (Blake, 2013).

The approach that I am using, which is the holistic approach, honors the inner wisdom of the body with its innate healing mechanisms and it recognizes that emotional healing is possibly even more important that physical cures. The holistic approach accepts both the Western and Eastern philosophies ans finds common ground in the areas that encourage the mind/body concepts, accepting the idea that mind is as much a part of health as is proper nutrition. Holism includes the body's physiological responses but does not exclude the emotions.

Holism incorporates the energy system of the body and sees stress factors being as real as infection. Holism focuses on maintaining the vitality of the organism and allows for the growth of the individual through empowerment. A holistic approach recognizes that the mind is capable of healing the body.

A beneficial offshoot of the holistic healing process occurs when a person integrates the hemispheres of the brain. As the mind and body are fully integrated with consciousness and subconsciousness, this process, known as horizontal brain integration, benefits certain physiological aspects of the body. Over time, it en-trains the neurological system, expanding conscious awareness. It seems that this process creates a never-ending circle of expansion and peace; it fully integrates the nervous system. But the first basis of chronic illness must be addressed-- which is stress.

Dr. Barbara Brown discusses the effects of stress and illness, "The condition becomes the diagnosis rather than the cause of the problem becoming the diagnosis". Dr. Brown explains that there is a known relationship between ill emotions and ill health.

From a holistic perspective, when observing health and wellness, all aspects of one's life becomes important, including mind, body and spirit. Each aspect of the human organism is vital, but, in understanding people, the scope of the various networks and inter-relationships of the body systems is too big to put your arms around it.

My goal is to understand how stress has impacted a person's health, as well as a person's physiological condition affecting the psychological condition, and creating a holistic framework that encompasses the conditions that are inter-related to the person's health, therefore, creating not only a natural medication that will help them, but also teaching and educating them on their condition so they know how to approach it, control it, and remain stable.

But as a concept, stress has been evaluated by the Eastern sciences and its casual relationships have been understood for years. Stress from an Eastern perspective is due to a mind that is in a continual state of unrest. It all begins with our thoughts. Thoughts are something of substance. This substance has the same quality of Schrodinger's wave packets (McEvoy 140) or the "bio-information" that is actively flowing through our bodies. Thought prints itself onto the body.

My Decompartmentalization Framework is a framework that I created and designed based on an holistic and integrative approach.

To Decompartmentalize means to remove excessive compartmentalization; to restore from a compartmentalized state; to merge back together.

In psychology, compartmentalization is defined as a defense mechanism where someone suppresses their thoughts and emotions. It is not always done consciously, but this can often justify or defend a person's level of engagement in certain behaviors.

Decompartmentalize- to organize something into departments

Compartmentalize- is to separate something into different categories

This is a great way to manage difficult parts of your life.

Compartmentalizing is unhealthy. Its primary a defense mechanism against psychological trauma but can also be used to block off disturbances or feelings, which, while needing to be dealt with at some time, are intrusive to the hypothetical current task.

The Decompartmentalization Framework: Transforming Health and Well-being for a Fulfilling Lifestyle

In today's fast-paced world, stressors and stagnant situations can take a toll on our overall health and well-being. However, by adopting the decompartmentalization framework, we can put these challenges to the side and focus on improving our lifestyle by 40% within the first 30 days. By detoxifying the mind, body, and soul, we can rediscover our true selves and prevent mental breakdowns caused by physical illness. In this article, we will explore how prioritizing self-care, decompressing unhealthy habits, situations, and relationships can lead to self-control and self-love.

1. Understanding the Decompartmentalization Framework:

   The decompartmentalization framework emphasizes the integration of various aspects of health and wellness, including physical, mental, emotional, and spiritual dimensions. By breaking down the barriers between these compartments and addressing them holistically, individuals can achieve a more balanced and fulfilling lifestyle.
2. Prioritizing Self-Care:

   Putting yourself first is crucial for overall well-being. By dedicating time to self-care activities such as exercise, meditation, and relaxation techniques, you can reduce stress levels and improve mental clarity. This self-investment allows you to better handle stressors and stagnant situations while nurturing a sense of self-control and love.
3. Detoxifying Mind, Body, and Soul:

   Detoxification is not limited to the physical body; it also involves cleansing the mind and soul. Engaging in activities like journaling, therapy, and practicing mindfulness helps release emotional baggage, negative thoughts, and toxic relationships. This process enables you to open your mind to your true self, thereby fostering personal growth and a deeper understanding of your inner desires.
4. Preventing Mental Breakdowns:

   Physical illness can often lead to mental breakdowns. By taking proactive steps to maintain good physical health through regular exercise, a balanced diet, and adequate sleep, you can reduce the risk of mental health issues. The decompartmentalization framework encourages individuals to prioritize their physical well-being as an integral part of their overall health.
5. Decompressing Unhealthy Habits, Situations, and Relationships:

To gain a sense of self-control and love, it's essential to identify and decompress unhealthy habits, situations, and relationships. This may involve setting boundaries, seeking support from loved ones, or making necessary lifestyle changes. By consciously letting go of detrimental influences, you create space for positive growth and a renewed sense of self.

The decompartmentalization framework offers a transformative approach to integrative health and medicine. By putting stressors and stagnant situations to the side and focusing on overall health and well-being, individuals can experience a 40% improvement in their lifestyle within the first 30 days. Through detoxifying the mind, body, and soul, one can rediscover their true self, prevent mental breakdowns, and gain a sense of self-control and love. Embracing this framework enables individuals to live a more fulfilling and balanced life, reaping the benefits of holistic health and wellness.

The Decompartmentalization Framework is An Integrative Approach to Overcoming Excessive Compartmentalization

In today's fast-paced world, managing various aspects of our lives can be challenging. We often find ourselves dividing our time, attention, and emotions into different compartments, which can lead to excessive compartmentalization. However, this approach can be unhealthy, hindering our overall well-being. In this article, we explore the decompartmentalization framework-a method that promotes an integrative approach to removing excessive compartmentalization and restoring balance in our lives.

Understanding Compartmentalization:

Compartmentalization is a common defense mechanism against psychological trauma or disturbances. It involves separating different aspects of our lives into distinct categories. While this may provide temporary relief from overwhelming emotions or intrusive thoughts, it can prevent us from addressing underlying issues and hinder personal growth.

The Drawbacks of Compartmentalization:

Compartmentalization, when used excessively, can have negative consequences. It limits our ability to deal with emotions effectively and can lead to increased stress levels. Moreover, it restricts our capacity to focus on the present moment and can impede our overall productivity and happiness.

Introducing the Decompartmentalization Framework:

The decompartmentalization framework encourages individuals to organize their lives into departments while promoting a healthy balance between them. It involves breaking down the barriers between various aspects of our lives and adopting an integrative approach to address challenges and enhance well-being.

Steps to Implement the Decompartmentalization Framework:

1. Self-Reflection: Begin by acknowledging the areas of your life that are excessively compartmentalized. Reflect on how this compartmentalization may be impacting your overall well-being.
2. Identify Priorities: Determine your priorities and values across different areas of your life, such as work, relationships, hobbies, and personal growth.
3. Find Synergies: Look for opportunities to integrate different aspects of your life. Seek connections and ways to combine activities or tasks that align with your priorities.
4. Establish Boundaries: While integrating various aspects of your life, it is essential to set clear boundaries to maintain balance and prevent overwhelm. Establish dedicated time for each department and honor those commitments.
5. Seek Support: Reach out to trusted friends, family members, or professionals who can provide guidance and support as you navigate the decompartmentalization process.

Benefits of Decompartmentalization:

By adopting the decompartmentalization framework, you can experience several benefits:

1. Enhanced Well-being: Decompartmentalization promotes a holistic approach to life, allowing you to address underlying issues and foster overall well-being.
2. Improved Focus and Productivity: By eliminating the mental barriers created by excessive compartmentalization, you can cultivate better focus and productivity in all areas of your life.
3. Authenticity and Emotional Growth: Decompartmentalization enables you to embrace your emotions fully and encourages personal growth by addressing emotional challenges head-on.

The decompartmentalization framework offers a valuable approach to remove excessive compartmentalization and restore balance in our lives. By integrating various aspects of our lives and addressing underlying issues, we can experience enhanced well-being, improved focus, and personal growth. Embracing this integrative approach can lead to a more fulfilling and connected life.

Also, Nutritional Medicine in Brain Development is important due to the fact that brain cells make neurotransmitters that act like signaling agents from one nerve cell to another (synaptic left), which are important in:

1. brain development
2. learning and memory
3. alertness and focused attention
4. arousal
5. sleep
6. mood
7. cognition
8. motivation and reward behavior

Norepinephrine is required for alertness, arousal and influences on the reward system. Decreased synthesis or release of norepinephrine is a common factor in ADHD, depression, and hypotension. Epinephrine is required for memory consolidation. Dopamine has many functions in the brain, including important roles in behavior and cognition, motivation and reward, sleep, mood, motivation, attention and learning.

A genetic defect in dopa-decarboxylase, or a deficiency in Vitamin B6 or magnesium can dramatically affect mental performance and behavior. However, high doses of Vitamin B6 can cause neurotoxicity, and must be monitored closely.

In the brain, serotonin plays an important role in the modulation of:

1. anger
2. aggression
3. mood- depression; which results from serotonin insufficiency. Sunlight increases serotonin levels as does amino acids found in foods and supplementation with 5-hydroxy-tryptophan. Serotonin is found in mushrooms and plants, including fruits and vegetables.

Most of the dry weight of the brain is lipids (fat). The outer skin (membrane) of brain cells require EFA's for nerve conduction (electrical impulses),and transmission from nerve to nerve. The brain likes access to omega-3 fats. The brain has higher levels of DHA levels than most other body tissues. However, deficiencies in omega-3 fats can impair brain development and function, affecting mental performance. Essential fatty acids are indispensable structural components of the cell membranes of all tissues.

The brain tries to maximize the efficiency of our thinking by recognizing familiar patterns and anticipating them when we look out into the world. Two systems in the brain mold out perceptions. On the other hand, there is the unconscious system that recognizes patterns, anticipates based on those patterns, and deduces how the perceptual fragments fit together. There is the conscious system that accepts the calculations of the unconscious-- questioning them when necessary-- and formulates decisions based on the wealth of background knowledge to which it has access.

The unconscious system in the brain pieces together fragments of our perceptions, anticipating patterns and filling in gaps when necessary, in order to devise a single, meaningful interpretation. It tells a story. The conscious system experiences that story but our can also reflect on it and even question it. The unconscious system in the brain is a straightforward logical system. When it detects seemingly irreconcilable stimuli, such as the feeling of someone being there when nobody's around, the brain generates the best story it can with the information at hand. It picks out the salient features of what we see and feel, scanning the depths of our memory, our beliefs, or hopes, and our worries to find patterns. It tries to concoct a satisfying explanation. It searches for meaning. By framing our perceptions in a unified narrative, the brain constructs the experience of life.

They feel separated from the world, distant from everyone around them, even the people they know most intimately. The Cotard delusion is a failure to connect perceptions with emotions. Neurologically, it's associated with a disconnect between 2 areas of the brain: the sensory system ad the limbic system. The limbic system processes emotions and memories and includes regions like the amygdala and the hypothalamus, which are located at the interior surface of the temporal lobe. When damage to the temporal and parietal lobes interrupts the communication between the sensory and the limbic system, the theory goes, patients will see, hear, and smell the world as they usually do but without having any emotional reactions.

The brain has a tendency to fill voids in our thinking and perceptions. Whenever they may be incomplete. Each time, the brain fills in the gaps; it does so with a purpose; to preserve our sense of self. The conscious system is thoroughly focused on protecting our personal narrative; the stability of human identity and its efforts are never more evident than the cases of emotional trauma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of anxiety, schizoaffective disorder, bipolar disorder, ADHD, Dementia, or other psychological issues and disorders; autoimmune disease such as fibromyalgia, lupus, and thyroid disease, neuropathy and chronic fatigue syndrome
* Must be able to swallow tablets

Exclusion Criteria:

* Children under the age of 18
* Must not be on any blood thinner medications
* Chronically ill patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-06-29 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Primary Outcomes for those diagnosed with Psychoneuromentalism Disorder | 4-6 weeks
  Memory will become more clear.

SECONDARY OUTCOMES:
Primary Outcomes for those diagnosed with Psychoneuromentalism Disorder | 8-12 weeks
  An improvement in mental health and psychological symptoms and functioning across various domains in life

OTHER OUTCOMES:
Primary Outcomes for those diagnosed with Psychoneuromentalism Disorder | 2-3 weeks
  Reduced Stress
Primary Outcomes for those diagnosed with Psychoneuromentalism Disorder | 6-8 weeks
  Reduced Anxiety Levels

CONTACTS AND LOCATIONS:
Overall Officials: Faith A Richardson, BSW, MPA, PhD, Study Director — Restored Purpose Counseling Alliance

IPD SHARING:
Plan to Share IPD: Yes
At this time, I don't have a specific plan set in place. I will take the necessary steps to make the IPD available to other researchers once I come up with a description.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will become available on January 7, 2023.
Access Criteria: Please send me an email if you would like to have access to my research and reports.
URL: https://www.hethforlifeholisticwellnesscenter.com